CLINICAL TRIAL: NCT06624345
Title: Inspiratory Training and Aerobic Exercise for Muscle Recovery in Myasthenia Gravis Post-Hospitalization
Brief Title: Interval Inspiratory Training and Aerobic Exercise for Muscle Recovery in Myasthenia Gravis Post-Hospitalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Collaborators: Chang Gung University of Science and Technology (Other); Kaohsiung Chang Gung Memorial Hospital,Taiwan (Unknown)
Responsible Party: Principal Investigator, Hui-Ling Lin, Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202002115A3
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Myasthenia Gravis
Keywords: myasthenia gravis; inspiratory muscle training; respiratory muscle strength; spirometery
MeSH Terms: conditions — Myasthenia Gravis | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory Muscle Training (Experimental): Subjects participated in a combination of inspiratory muscle training and aerobic exercise for approximately 30 minutes per day over a period of six weeks.
  Interventions: Procedure: Inspiratory muscle training
- Control group (Sham Comparator): Subjects received routine care.
  Interventions: Procedure: Control Group

INTERVENTIONS:
Procedure: Inspiratory muscle training — Patients in the IMT group received the intervention using a threshold loading device set at a pressure range of 5-39 cmH₂O. They were instructed to perform six sets of five breaths, totaling 30 breaths, twice daily for six weeks. Additionally, the aerobic exercise regimen included upper limb exercises (raising arms without resistance), a lower limb stepping warm-up, and a walking routine consisting of 5 minutes of slow walking, 2 minutes of brisk walking, and another 5 minutes of slow walking, for a total of 30 minutes per day.
  Arms: Inspiratory Muscle Training
Procedure: Control Group — Subjects received routine care.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to determine whether inspiratory muscle training aids in the recovery of respiratory muscle strength and helps prevent further muscle weakness in patients with myasthenia gravis.

The primary research questions are:

Does inspiratory muscle training enhance respiratory muscle strength recovery? Does the intervention lead to improved lung volumes? Participants underwent daily inspiratory muscle training and aerobic exercise for six consecutive weeks.

DETAILED DESCRIPTION:
Patients with myasthenia gravis who experience acute exacerbations requiring hospitalization often suffer a significant decline in muscle strength, followed by partial recovery after the acute phase. This randomized controlled trial aims to evaluate the potential of early inspiratory muscle training and aerobic exercise in promoting muscle strength recovery and preventing further weakness. The study will assess differences in lung function, respiratory muscle strength, and dyspnea levels following the intervention after patients are discharged from the hospital post-acute exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized due to a myasthenia gravis crisis
* Cleared for discharge from the hospital
* Capable of completing six weeks of home-based respiratory muscle and exercise training

Exclusion Criteria:

* Myasthenia Gravis Foundation of America (MGFA) classification I or V
* Presence of concurrent heart, kidney, liver, or metabolic diseases, or malignant tumors
* Ability to follow exercise instructions
* New York Heart Association (NYHA) Class III/IV
* Pulmonary disease (FEV1/FVC ratio < 0.7 and FEV1 < 50% predicted)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum inspiratory pressure | Six weeks
  Maximum inspiratory pressure was measured by instructing each subject to exert their maximum inspiratory force against a pressure gauge.

SECONDARY OUTCOMES:
Dyspnea Severity Assessment | Six weeks
  Dyspnea severity was assessed by a rating of perceived exertion, using the Borg Scale which ranged from 0 (no respiratory difficulty) to 10 (extreme respiratory difficulty), with higher scores indicating more severe breathing difficulty.
Forced expiratory volume at one second | Six weeks
  The forced expiratory volume at one second was obtained, using spirometry, by having the patient take a deep breath and then exhale forcefully. The test results were based on three reproducible measurements.
Peak expiratory flow | Six weeks
  The peak expiratory flow was measured using a respiratory mechanics monitor during three forceful expirations.
Maximum expiratory pressure | Six weeks
  Maximum expiratory pressure was measured by instructing each subject to exert their maximum expiratory force against a pressure gauge.
Forced Vital Capacity | Six weeks
  Forced vital capacity was measured using spirometry. Patients were instructed to take a deep breath and then exhale forcefully. The results were based on the average of three reproducible measurements.
Six-minute walk test | Six weeks
  Patients were instructed to walk as fast as possible, while pulse oxygen saturation levels, heart rate, and Borg scale scores were monitored and recorded before, during, and after the test.

CONTACTS AND LOCATIONS:
Overall Officials: Jui-Fang Liu, PhD, Principal Investigator — Chang Gung University of Science and Technology
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The data is available upon request from the principal investigator.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available 3 years after the registration
Access Criteria: The data is available upon request from the principal investigator.

REFERENCES:
- [Derived] Chang CL, Fang TP, Tsai HM, Chen HC, Liu SF, Lin HL, Liu JF. Inspiratory muscle training and aerobic exercise for respiratory muscle strength in myasthenia gravis post-hospitalization- a randomized controlled trial. BMC Pulm Med. 2025 May 27;25(1):266. doi: 10.1186/s12890-025-03733-7. PMID 40426137